CLINICAL TRIAL: NCT00915187
Title: A Phase II Safety and Immunogenicity Study of Intramuscular CCS/C-adjuvanted Influenza Vaccine in Elderly, a Double-blind Randomized, Controlled Single Center Study
Brief Title: Safety and Immunogenicity Study of Intramuscular CCS/C-adjuvanted Influenza Vaccine in Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NasVax Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NX09-4
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Influenza
Keywords: Vaccination, influenza prevention
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator)
  Interventions: Biological: Influenza Vaccine
- CCS/C (Adjuvant Formulation) (Experimental)
  Interventions: Drug: CCS/C

INTERVENTIONS:
Drug: CCS/C — Adjuvant to influenza vaccine
  Arms: CCS/C (Adjuvant Formulation)
Biological: Influenza Vaccine — Influenza vaccine
  Arms: Control

SUMMARY:
To examine the safety and immunogenicity of two formulation of liposomal adjuvant / delivery system (VaxiSomeTM=CCS-Cholesterol [CCS/C]), combined with commercial influenza vaccine in an elderly healthy population when given once intramuscularly (IM).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older, mentally competent, willing and able to give written informed consent prior to study entry, male or female;
* able to comply with all the study requirements;
* in stable good health as determined by medical history; physical examination; clinical judgment of the investigator.
* Have adequate renal function (renal clearance of at > 30ml/min)
* Have normal liver function (hepatic transaminases [ALT and AST] < 43 U/L)
* Have hemoglobin > 11.5 g/L

Exclusion Criteria:

* Any serious chronic or acute disease (in the judgment of the investigator) including but not limited to: cancer, except for localized skin cancer;
* Advanced congestive heart failure; Acute exacerbation of Chronic obstructive pulmonary disease (COPD); Autoimmune disease, Acute or progressive hepatic disease; Acute or progressive renal disease with a renal clearance of at < 30ml/min ; Severe neurological or psychiatric disorder; History of Guillain Barré syndrome; Severe asthma.
* Clinically significant symptoms of neurological disease; untreated hypertension; increased liver enzymes.
* History of any anaphylactic reaction and/or serious allergic reaction following a vaccination

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Immunogenicity will be evaluated according to the CHMP criteria for evaluation of flu vaccines, i.e., Seroprotection, Geometric Mean Ratios, and Seroconversion rate | Day 28 following vaccination

SECONDARY OUTCOMES:
Immunogenicity will be evaluated according to the CHMP criteria for evaluation of flu vaccines, i.e., Seroprotection, Geometric Mean Ratios, and Seroconversion rate | Day 90 following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Clinical Pharmacology Unit, Division of Medicine, Hadassah University Hospital Jerusalem, Israel
Locations (1):
- Clinical Pharmacology Unit, Division of Medicine, Hadassah University Hospital, Jerusalem, Israel